CLINICAL TRIAL: NCT07011771
Title: A Phase 1/2 Dose-Escalation Trial to Evaluate Safety, Tolerability, and Efficacy of a Single Dose of CAP-003 Gene Therapy Administered to Patients With Parkinson's Disease With GBA1 Gene Mutation (PD-GBA)
Brief Title: A Clinical Trial of CAP-003 Gene Therapy in Adult Patients With GBA1 Associated Parkinson's Disease
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per protocol stopping rule was met for a separate trial for a different disease state and different experimental therapy that utilized a similar technology.
Sponsor: Capsida Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAP-003-101
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: GBA1 Parkinson Disease
Keywords: GBA1; Gene Therapy; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Level 1 (Experimental): Participants will receive a single dose of CAP-003, administered IV
  Interventions: Drug: gene therapy
- Dose Level 2 (Experimental): Participants will receive a single dose of CAP-003, administered IV
  Interventions: Drug: gene therapy

INTERVENTIONS:
Drug: gene therapy — IV gene therapy
  Arms: Dose Level 1
Drug: gene therapy — IV gene therapy
  Arms: Dose Level 2

SUMMARY:
The goal of this clinical trial is to learn about the safety of CAP-003 gene therapy in adults with GBA1 associated Parkinson's Disease. It will also provide information about whether CAP-003 demonstrates efficacy in these adults.

Participants will have a single intravenous infusion of CAP-003 and visit the clinic regularly for 2 years for checkups and tests.

DETAILED DESCRIPTION:
This is a Phase 1/2, first-in-human, open-label, multi-centre, dose escalation trial to assess the safety, tolerability, and efficacy of a single intravenous (IV) dose of CAP-003 administered to adult patients aged 21 to 75 with Parkinson's Disease associated with GBA1 mutation.

Approximately 31 participants will be dosed in this trial. Phase 1 is a dose escalation phase that will dose approximately 6 participants divided into 2 cohorts (Cohort 1 and Cohort 2) while Phase 2 will have 1 dose cohort and dose approximately 25 participants. Participants in Phase 1 will be dosed sequentially in each cohort. Phase 2 will allow participants to be dosed concurrently if safety and tolerability data from Phase 1 are deemed acceptable.

Participants will receive a single IV infusion of CAP-003 and will then be followed for 2 years with safety measures, assessments to measure changes from Baseline in motor and non-motor scales, cognitive function, patient and clinical global impression of severity and improvement, disease progression, sleep scale and suicide severity rating.

Upon completion of the study or at the participant's final visit they will be invited to participate in a 3 year safety follow up study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21 to 75 years
* Has diagnosis of Parkinson's disease (PD) per UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria;
* Has modified Hoehn and Yahr Stage I to III in the 'OFF' state;
* Presence of a pathogenic or likely pathogenic GBA1 mutation confirmed;
* Must be generally ambulatory, not dependent on wheelchair;
* Has a body weight of ≥40 kg (88 lb) to ≤110 kg (242 lb) and a body mass index (BMI) of 18 to 34 kg/m2;
* Participant has a reliable study partner/informant (eg, family member, friend) willing and able to participate in the trial as a source of information on the participant's health status and cognitive and functional abilities;
* Is living in the community (ie not in a nursing home)

Exclusion Criteria:

* Presence of a bi-allelic GBA1 mutation, or presence of LRRK2 2019S or other LRRK2 mutation;
* Diagnosis of significant central nervous system (CNS) disease other than PD that may be a cause for the participant's PD symptoms or may confound study objectives;
* Montreal Cognitive Assessment (MoCA) score of ≤22;
* History of deep brain stimulator placement, focused ultrasound therapy, or other intercranial surgery for PD;
* Hypersensitivity or contraindications to corticosteroid;
* Prior gene or cell therapy;
* Positive test result for anti-capsid total antibodies (tAb);
* Unable to undergo lumbar puncture;
* Diagnosis of Gaucher disease;
* Clinically significant abnormalities in safety lab tests, vital signs;
* Other illnesses or medications that may affect the interpretation of the study results.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) | 2 years
  Incidence of treatment emergent adverse events assessed through clinical safety laboratory tests (hematology, chemistry, liver function and urinalysis), ECG, vital sign measurements and physical examinations

SECONDARY OUTCOMES:
Efficacy: Glucosylsphingosine (GluSph) biomarker change | Baseline, week 4, week 8, week 12, month 6, month 12, month 18, month 24 or end of trial
  Percent change from baseline in GluSph levels in plasma. Higher percent decrease is a better outcome.
Efficacy: Glucosylsphingosine (GluSph) biomarker change | Baseline, week 12, month 6, month 18
  Percent change from baseline in GluSph levels in CSF. Higher percent decrease is a better outcome.
Efficacy: β-Glucocerebrosidase (GCase) biomarker change | Baseline, week 4, week 8, week 12, month 6, month 12, month 18, month 24 or end of trial
  Percent change from baseline in GCase protein levels in plasma. Higher percent increase is a better outcome.
Efficacy: β-Glucocerebrosidase (GCase) biomarker change | Baseline, week 12, month 6, month 18
  Percent change from baseline in GCase protein levels in CSF and plasma. Higher percent increase is a better outcome.
Efficacy: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) disease rating change | Baseline, month 6, month 12, month 18, month 24 or end of trial
  Change from baseline in MDS-UPDRS Parts II and III. A decrease in score indicates improvement of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Brandabur, MD, Study Director — Capsida Biotherapeutics
Locations (6):
- United States (6):
  - Rush University Medical Center, Chicago, Illinois
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Booth Gardner Parkinson's Care Center - Evergreen Neuroscience Institute, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No